CLINICAL TRIAL: NCT03299855
Title: MoCA vs. MMS: Which Tool to Detect Cognitive Disorders in Oncogeriatric?
Acronym: MOCA-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: UCOG (Unite de coordination en Onco-Gériatrie) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 2017-A01079-44
Record Dates: First submitted 2017-09-26; First posted 2017-10-03 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-09

CONDITIONS: Neoplasms
Keywords: oncogeriatric; MMS; MoCA
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Passation of MMS and MoCA tests associated to passation of neuropsychological test
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Passation of neuropsychological test — Passation of MoCA and MMS tests associated with neuropsychological test

SUMMARY:
This study concerns elderly patients with cancer with onco-geriatric assessment.

This study propose to associate the collection of the results with the Mini-Cog and the CODEX with the passing of the MoCA and the MMS tests, as well as a neuropsychological assessment, in order to determine if the patients have cognitive impairments, to evaluate the sensitivity of these 4 screening tests in elderly patients seeking treatment for their cancer. The results of this study will make it possible, where appropriate, to adapt the practice in the context of oncogeriatric assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 70 years
* Patient with cancer (solid tumor or haemopathy) for whom a first line treatment is envisaged (whatever it is). Surgery and radiotherapy are allowed before entry into the study.
* Patient candidate for oncogeriatric assessment
* Patient agree to participate in the study
* Using the French language

Exclusion Criteria:

* Primary central nervous system or cerebral metastasis
* Evolutionary psychiatric pathology known (e.g. schizophrenia)
* Severe Visual and / or Auditory Impairment
* Patients unable to respond to cognitive tests
* Patient (s) deprived of liberty, under guardianship or curatorship
* Refusal of participation

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 104 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
Evaluate the sensitivity of MoCA test | Up 2 months after inclusion, before initiation of treatment
  MoCA is considered clinically relevant if its sensitivity to identify patients with cognitive impairment is at least 75%

CONTACTS AND LOCATIONS:
Overall Officials: florence JOLY, prof, Principal Investigator — Centre François Baclesse
Locations (6):
- France (6):
  - Centre François Baclesse, Caen
  - CHU, Caen
  - CH, Cherbourg
  - Ch Compiegne, Compiègne
  - Centre Henri Becquerel, Rouen
  - Centre Hospitalier, Saint-Lô

IPD SHARING:
Plan to Share IPD: No